CLINICAL TRIAL: NCT02432534
Title: Atorvastatin in Active Vitiligo: a Bicentric Prospective Randomized Trial
Brief Title: Atorvastatin in Active Vitiligo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-AOI-01
Record Dates: First submitted 2015-04-10; First posted 2015-05-04 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2017-03

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- UVB + treatement (Experimental): The patients will be treated with the combination of oral atorvastatin and NBUVB phototherapy twice a week for 6 months.
  Interventions: Drug: Atorvastatin
- UVB (Other): The patients will be receiving only NB-UVB phototherapy twice a week for 6 months.
  Interventions: Other: UVB

INTERVENTIONS:
Drug: Atorvastatin — The patients will be treated with the combination of oral atorvastatin and NBUVB phototherapy twice a week for 6 months. The initial starting dose of the oral atorvastatin will be 40mg daily and after 1 month, if tolerated clinically and biologically following blood tests, the dose will be increased to 80mg daily.
  Other Names: UVB
  Arms: UVB + treatement
Other: UVB — The patients will be receiving only NB-UVB phototherapy twice a week for 6 months.
  Arms: UVB

SUMMARY:
Condition:

Non segmental and active vitiligo of adulthood.

Main objective:

To evaluate the efficacy of a daily treatment with atorvastatin 80mg/d combined to UVB compared to UVB alone in active vitiligo after 6 months of treatment.

Methods:

Prospective interventional bicentric study with evaluation blinded to the treatment received.

Inclusion criteria:

Patients from 18 to 75 year-old with active non segmental vitiligo. Active is defined by the apparition or the modification of vitiligo lesions with the past 3 months and under Wood's lamp examination hypochromic borders and/or spotty depigmentation.

Interventions:

After central randomization

* Arm A : atorvastatin 40mg/d for 1 months then 80mg/d for 5 months combined with twice weekly narrowband UVB treatment for 6 months.
* Arm B: with twice weekly narrowband UVB treatment for 6 months.

Evaluation:

Main criteria: Decrease of VASI score expressed in percentage Secondary criteria: Decrease of VETF score expressed in percentage. Variation of PGA and DLQI scores. Clinical and biological tolerance. Variation of CXCL10 levels in the serum.

Length of the study:

Inclusion period: 12 months. Length of treatment: 6 months. Statistical analyses and drafting the article: 6 months. Total length: 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Active non-segmental vitiligo defined by

  * Non- segmental vitiligo with new patches or extension of old lesions during the last 3 months AND
  * Presence of hypochromic aspect under Wood's lamp examination and/or perifollicular hypopigmentation under Wood's lamp examination
* Patient requiring a treatment by UVB
* Signed informed consent document
* Patient registered to the French Social Security

Exclusion Criteria:

* - Segmental or mixed vitiligo
* Pregnant (urinary pregnancy test will be done) or lactating patients
* Allergy to statin medications
* Use of statin or fibrate medications due to cardiac risks
* Use of statin medications in the past 8 weeks
* Use of any medications contraindicated with use of statin medications
* Use of vitiligo treatments (both topicals and phototherapy) in the past 4 weeks
* Treatment with immunomodulating oral medications in the past 4 weeks
* Hepatic disease and/or dysfunction
* Renal dysfunction
* Personal or familial history of myopathy or personal history of rhabdomyolysis or elevated baseline creatinine kinase
* Alcohol or drug abuse
* Untreated hypothyroidism
* Personal history of skin cancer
* Any other clinically significant findings that, in the opinion of the Principal Investigator, might interfere with study evaluations or pose a risk to subject safety during the study.
* Patients assessed to be uncooperative
* Participants in other clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Percentage of decrease in Vitiligo Area Scoring Index (VASI) score | 4 times (baseline, 1 month, 3 month and 6 month)
  Percentage of decrease in Vitiligo Area Scoring Index (VASI) score between baseline and 6 months after commencement of the study. In the VASI assessment, the body is separated into five sites: hands, upper extremities, trunk, lower extremities and feet. The extent of residual depigmentation is expressed by the following percentages: 0, 10%, 25%, 50%, 75%, 90%, or 100%. The VASI score is then derived by multiplying the values assessed for the vitiligo involvement by the percentage of affected skin for each body site and summing the surface of the lesions of all body sites together.

SECONDARY OUTCOMES:
VETF | 4 times (baseline, 1 month, 3 month and 6 month)
  Percentage of decrease in Vitiligo European Task Score (VETF) score between baseline and 6 months after commencement of the study.
PGA | 4 times (baseline, 1 month, 3 month and 6 month)
  Physician global assessment (PGA). Treatment response will be graded as excellent (76 - 100%), moderate (51 - 75%), Mild (26 - 50%), minimal (1 - 25%) or no response.
Adverse event | 4 times (baseline, 1 month, 3 month and 6 month)
  Description of potential side effects using clinical evaluation and biology. Clinical and biological tolerability of high dose of oral atorvastatin will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice; Chuah Sai Yee, Ph, Principal Investigator — Singapour
Locations (2):
- CHU de Nice, Nice, Alpes-Maritimes, France
- National Skin center - 1 Mandalay Rd, Bedok, Singapore, Indonesia